CLINICAL TRIAL: NCT00826345
Title: Patient-Oriented TCM Intervention for DSP in HIV: A Pilot Study
Brief Title: Acupuncture/Moxibustion (Acu/Moxa) for Distal Symmetric Peripheral Neuropathy (DSP) in HIV
Acronym: TCMAcuPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Joyce Anastasi, Professor / Director Div. Special Studies in Symptom Management, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAD3398
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Peripheral Neuropathy; HIV; AIDS; HIV Infections
Keywords: Peripheral Neuropathy; Neuropathy; HIV; AIDS; DSP; alternative therapies
MeSH Terms: conditions — Peripheral Nervous System Diseases; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture/Moxibustion (Experimental): Diagnostic Acupuncturists assessments will inform acupuncture/moxibustion treatment prescriptions for persons with HIV/AIDS experiencing distal peripheral neuropathy. This protocol is tailored specifically for the subject's unique diagnosis according to the symptoms being reported at each diagnostic acupuncture (DA) session.
  Interventions: Other: Acupuncture / Moxibustion
- Placebo Acupuncture / Moxibustion (Placebo Comparator): Sham/placebo Arm: Points will be administered away from the classic/traditional true point location.
  Interventions: Other: Acupuncture/Moxibustion

INTERVENTIONS:
Other: Acupuncture / Moxibustion — Acupuncture/Moxibustion points will be administered per point prescription.
  - Active
  Arms: Acupuncture/Moxibustion
Other: Acupuncture/Moxibustion — Sham/Placebo Acupuncture/Moxibustion - Not active
  Arms: Placebo Acupuncture / Moxibustion

SUMMARY:
This preliminary study will investigate the use of Acupuncture and Moxibustion (Acu/Moxa) for distal symmetric peripheral neuropathy (DSP) associated with HIV applying traditional Chinese medicine (TCM) evaluations conducted by a diagnostic acupuncturist. The investigators will evaluate the role of Acu/Moxa in reducing the symptoms of DSP related to HIV/AIDS and treatment side effects. The effects of symptom reduction on quality of life will also be examined. This application will establish a proof of principle for the role of Acu/Moxa in the treatment of DSP and provide data that will serve as a foundation for establishing a future larger clinical trial.

DETAILED DESCRIPTION:
This study is a prospective, randomized, sham/placebo controlled, blinded (subject and evaluator), parallel groups clinical trial. This preliminary study will investigate the use of Acupuncture and Moxibustion (Acu/Moxa) for DSP associated with HIV applying TCM evaluations conducted by a diagnostic acupuncturist. The investigators will evaluate the role of Acu/Moxa in reducing the symptoms of DSP related to HIV/AIDS and treatment side effects. The effects of symptom reduction on quality of life will also be examined. Data from daily symptom diaries and questionnaires will be analyzed with mixed model analysis of variance for between group difference in the temporal pattern of symptom reduction at baseline, after 6 weeks of twice weekly treatment, and after a no-treatment follow-up session. In addition, exploratory analyses will assess the logistics of a CAM clinical trial for HIV/AIDS related DSP in preparation of a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women HIV positive or CDC defined AIDS diagnosed subjects who are 18 years of age or older, have a history of distal symmetrical peripheral neuropathy of the lower extremities (legs and feet) for two months or greater.
* Experiencing patient rated pain severity at "moderate" on the Gracely pain scale documented in 1 week prospective self report symptom diary.
* Verification from Primary provider of subject's: HIV status, diagnosis of DSP, and their agreement that their patient is clinically suitable for the study.
* Individuals able to successfully complete a mini-mental status exam (obtaining a score of 24 or above).
* Individuals who understand and agree to complete daily symptom diaries for the duration of the study.
* Individuals taking antiretroviral combinations (a) must have completed an initial 8 weeks of a stable regime (same drug(s), dose & frequency) prior to entry into the study.
* Individuals taking chronic pain medications (b) must be on a stable regime (same drug, dose & frequency) for at least twenty one (21) days prior to entry into the study.
* Individuals on all other medications which may have neuropathy listed as a side effect must be on a stable regime (same drug(s), dose & frequency) for at least 21 days prior to entry in the study.

Exclusion Criteria:

* Individuals with an acute medical condition, i.e. pneumocystis carinii pneumonia, tuberculosis and or other opportunistic infections or conditions that would require medical attention.
* Individuals with diagnosis of diabetes mellitus, B12 deficiency
* Topically applied medications to the lower extremities.
* Individuals with alcohol and/or substance dependence.
* Individuals with bleeding tendency
* Currently receiving treatment with corticosteroids
* Use of INH, dapsone or metronidazole within 8 weeks prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Symptom diary Gracely Pain Scale | Baseline, Weekly and Follow-up visits

SECONDARY OUTCOMES:
Subjective Peripheral Neuropathy Screen (SPNS) Clinical Global Impression Scale Neurological Assessment Form | Baseline, weekly and follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Anastasi, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States